CLINICAL TRIAL: NCT06308250
Title: Comparative Effects of Mime Therapy and Action Observation Therapy on Facial Symmetry and Quality of Life in Bell's Palsy
Brief Title: Comparative Effects of Mime Therapy and Action Observation Therapy in Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0294
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Bell Palsy
Keywords: Bell Palsy; Breathing exercise; Comparative; MIME Protocol; Randomized clinical trial
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A ( MIME THERAPY) (Experimental): Group A will receive mime therapy of 30 minutes with short resting intervals. Treatment will be given 5 times per week for 6 weeks. Mime therapy consist of:
  1. Self massage of 10 minutes,
  2. Breathing and relaxation exercises of 5 minutes,
  3. Articulation of 5 minutes and
  4. Facial expression exercises of 10 minutes.
  Interventions: Other: MIME THERAPY
- GROUP B (ACTION OBSERVATION THERAPY) (Experimental): Group B will receive action observation therapy of 30 minutes with short resting interval. The treatment will be given 5 times per week for 6 weeks.
  During the presentation of a video clip, patients sit relaxed in front of the computer screen while observing it.
  After observing a motor act for 3 min (observation phase) patients are required to imitate what they observed for 2 min (execution phase).
  Interventions: Other: ACTION OBSERVATION THERAPY

INTERVENTIONS:
Other: MIME THERAPY — Mime therapy consist of:
  Self massage: patients will be taught to massage their face and neck daily for about 10 minutes which includes effleurage and kneading of both sides of face.
  Breathing exercises: patient will be taught to recognize tension and feel the difference between tension and relaxation in facial musculature for 5 minutes. Expiration exercises will be used to induce relaxation.
  Articulation: vowels such as a,e,i,o,u and consonants such as p and b will be used to teach position of the lips for 5 minutes.
  Facial expression exercises: forehead wrinkle, smiling, eye closure, frowning, disgust, surprise, anger, sadness will be performed for 10 minutes
  Arms: GROUP A ( MIME THERAPY)
Other: ACTION OBSERVATION THERAPY — Function of each of the muscle is observed for 3 minutes and then executed for 2 minutes.
  Frontalis (Raising eyebrows and forehead wrinkling). Corrugator Supercili (Moving the eyebrow down and inward toward the nose and inner eye).
  Orbicularis oculi (Closing the eyelids). Buccinator (Blowing air in and out of the mouth). Zygomaticus major (Smiling). Orbicularis oris (Lip pursing or puckering).
  Arms: GROUP B (ACTION OBSERVATION THERAPY)

SUMMARY:
The aim of this study is to determine comparative effects of mime therapy and action observation therapy on facial symmetry and quality of life in Bell's palsy. Bell's palsy is characterized as an abrupt paralysis of the peripheral facial nerve, typically without a known cause. Mime Therapy is a performing technique that helps patients regain the ability to use their face muscles. Action observation therapy is novel rehabilitation approach exploiting this mirror mechanism.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Sir Ganga Ram Hospital in 7 months. 62 participants with Bell's palsy will be included as per sample size calculation through convenience sampling technique. Participants which meet inclusion criteria will be randomly allocated using online randomization tool into two groups. Group A will receive Mime therapy for 30 minutes with short resting interval and Group B will receive action observation therapy for 30 minutes. Each group will receive treatment session of 5 days per week for 6 weeks.

Facial symmetry will be measured using the 13-item Sunny Brook facial Grading System, Facial disability index will be used to assess the quality of life and The House-Brackmann Facial Nerve Grading System will be used to characterize the degree of facial paralysis. The data will be analyzed using SPSS version 24 for Windows software.

ELIGIBILITY:
Inclusion Criteria:

1. Bell's Palsy with acute onset of 1-3 weeks.
2. Unilateral loss of facial weakness.
3. Patients with intact taste sensation.
4. Bell's Palsy of House Brackmann grade 3 and 4.
5. Idiopathic Bell's Palsy.

Exclusion Criteria:

1. History of facial palsy recurrence.
2. Stroke associated Bells palsy.
3. History of pregnancy
4. Subjects with any disability, fracture, or tumor.
5. History of facial surgery.
6. Subject having skin allergy on face.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Sunny Brook Facial Grading System | 6th week
  The system includes three components: resting symmetry, the symmetry of voluntary movements, and synkinesis. A composite facial symmetry score is calculated as [4 × symmetry of voluntary movement - 5 × resting asymmetry + 1 × synkinesis] with 100 representing normal facial symmetry.
Facial Disability Index | 6th week
  it is used to assess the quality of life in patients with bell's palsy. It also helps to measure the difficulties of the face in activities of daily living. It represents the relationship between impairments, disability, and psychosocial status and also focuses on the disability of individuals with disorders of the facial motor system. The individual subscales are scored out of a total of 100 where the highest score is the best result.

CONTACTS AND LOCATIONS:
Overall Officials: Muhmmad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No